CLINICAL TRIAL: NCT04240106
Title: Multicenter,Open-label,Phase II Clinical Trial to Evaluate the Efficacy and Safety of Niraparib + Aromatase Inhibitors for(HR)+/(HER2)-, MBC With Either Germline BRCA-mutated or Germinal BRCA-wildtype and Homologous Recombination Deficiency
Brief Title: Niraparib Plus Aromatase Inhibitors for Luminal-like(HER2-,ER+) and gBRCA or HDR+ Metastatic Breast Cancer (LUZERN)
Acronym: LUZERN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP190; 2017-004323-72 (EudraCT Number)
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Breast Cancer Metastatic
Keywords: BRCA mutations; homologous recombination deficiency; Luminal like
MeSH Terms: conditions — Breast Neoplasms | interventions — niraparib; Aromatase Inhibitors

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, single-arm, two-cohort, Simon's two- stage phase II clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niraparib in combination with Aromatase Inhibitors (Experimental): Upon meeting all selection criteria, patients enrolled in the study will receive the combination of niraparib orally, once daily, flat- fixed, continuously in 28-day cycles plus aromatase Inhibitors.
  Interventions: Drug: Niraparib; Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Niraparib — Niraparib orally daily beginning on Day 1 and continuing through Day 28 of every 28-day cycle.
  Other Names: ZEJULA
Drug: Aromatase Inhibitors — Aromatase Inhibitors beginning on Day 1 and continuing through Day 28 of every 28-day cycle.

SUMMARY:
This study evalues the efficacy -as determined by the clinical benefit rate (CBR)- of niraparib in combination with AIs in unresectable locally advanced or metastatic HR-positive/HER2-negative breast cancer patients harboring either gBRCAms or gBRCAwt and HRD.

The planned number of patients is 23.

Investigational product is Niraparib and will be administered daily continuously in 28-day cycles plus aromatase Inhibitors.

Total study duration is 36 months and until 5 years of follow up.

DETAILED DESCRIPTION:
This is a Multicenter, Open-label, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Niraparib plus Aromatase Inhibitors for Hormone Receptor (HR)-positive/Human Epidermal Growth Factor Receptor 2 (HER2)-negative Metastatic Breast Cancers with either Germline BRCA-mutated or Germinal BRCA-wild-type and Homologous Recombination Deficiency (HRD).

The main objetive is to assess the efficacy -as determined by the clinical benefit rate (CBR)- of niraparib in combination with AIs in unresectable locally advanced or metastatic HR-positive/HER2-negative breast cancer patients harboring either gBRCAms or gBRCAwt and HRD.

Upon meeting all selection criteria, patients enrolled in the study will receive the combination of niraparib orally (according to baseline criteria described in Table 4), once daily, flat- fixed, continuously in 28-day cycles and AI that must be identical to the last AI-containing regimen.

A total of 23 patients will be recruited as follows:

* Stage I: N=6 patients in the cohort A;
* Stage II: N=8 patients in the cohort A; N=9 patients in the exploratory cohort B

The total duration of the study period is 36 months follow until 5 years of follow up.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients have been informed about the nature of study, including the exploratory sub-study and has agreed to participate and signed the informed consent prior to participation in any study related activities.
* 2. Male or female patients ≥ 18 years of age.
* 3. Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1 which the Investigator believes is stable at the time of screening.
* 4. Life expectancy ≥16 weeks.
* 5. Patients have a histologically and/or cytologically confirmed diagnosis of breast cancer.
* 6. Patients have radiologic evidence of inoperable locally recurrent or metastatic breast cancer (MBC) that are not candidates for curative intent.
* 7. Patients have human epidermal growth factor receptor 2 (HER2)- negative breast cancer (based on most recently analyzed biopsy) defined as a negative in situ hybridization (ISH) test or an immunohistochemistry (IHC) status of 0, 1+, or 2+ (if IHC 2+, a negative ISH test is required) by local laboratory testing.
* 8. Patients have hormone receptor (HR)-positive breast cancer (based on most recently analyzed biopsy) defined as estrogen receptor (ER) and/or progesterone receptor (PgR) with ≥10% of tumor cells positive for ER and/or PgR by IHC irrespective of staining intensity.
* 9. [Cohort A]: Patients with documented germinal mutation in BRCA1 or BRCA2 genes that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function). Patients with germinal mutations in BRCA1 or BRCA2 genes (gBRCAms) that are considered to be nondetrimental (e.g., "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favor polymorphism" or "benign polymorphism," etc.) will not be eligible for the study. Germinal BRCA1/2 results preceding the ICF signature will be accepted, as long as the results are documented and captured in the medical record during the pre-screening period.
* 10. [Exploratory cohort B]: : Patients with either germinal BRCA1/2 wild-type (gBRCAwt) or gBRCAms that are considered to be nondetrimental (e.g., "Variants of uncertain clinical significance" or "Variant of unknown significance" or "Variant, favor polymorphism" or "benign polymorphism," etc.) and homologous recombination deficiency (HRD) based on the Myriad myChoice® CDx PLUS test. HRD status will be centrally confirmed both on the most recent tumor tissue since last progression (from either metastasis or primary tumor) and blood samples. Patients with a Myriad myChoice® CDx PLUS score of ≥ 25 or greater will be considered to have an abnormal HRR pathway and defined as HRD.
* 11. [Exploratory cohort B]: Willingness and ability to provide additional six formalin-fixed paraffin-embedded (FFPE) tissue slides from the most recent tumor tissue since last progression (from either metastasis or primary tumor) to centrally perform the assay. It is strongly recommended obtaining six consecutive sections from the same tissue block used for the determination of HRD status.
* 12. At least one and up to two prior lines of endocrine therapy (aromatase inhibitors [AIs] or fulvestrant) for treatment of locally recurrent and/or metastatic disease (except for patients progressing in the neoadjuvant or adjuvant setting).
* 13. Confirmed disease progression while in the last AI-containing regimen (not necessarily in the treatment line immediately prior to study entry) with secondary endocrine resistance criteria.
* 14. Patients may have progressed on no more than one chemotherapy regimens in the metastatic setting.
* 15. The following will not be counted as a prior line of cytotoxic chemotherapy:

  * Prior hormonal therapy and non-hormonal targeted therapy.
  * Targeted and biologic therapies.
  * The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as this was started at least 5 days prior to study treatment.
* 16. Prior carboplatin- or other platinum compound-based therapy is allowed if have been administered in one of the following settings:

  * Disease-free interval > 12 months from date of completion of neoadjuvant or adjuvant treatment.
  * As potentially curative treatment for a prior non-breast cancer with no evidence of disease for ≥ 5 years.
* 17. Patients must have evaluable or measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1. Patient with bone-only metastases are eligible.
* 18. Willingness and ability to provide the most recent tumor biopsy since last progression from either metastatic or primary tissues both at the time of the inclusion and at disease progression or study termination in order to perform exploratory studies. If not feasible, patient eligibility should be evaluated by a Sponsor's qualified designee.
* 19. Patients must agree to provide blood samples at the time of study inclusion, every three cycles of treatment, and upon disease progression or study termination in order to perform exploratory studies.
* 20. Adequate hematologic and organ function within 28 days before the first study treatment on Cycle 1 Day 1.
* 21. Female patients of childbearing potential must have a negative serum pregnancy test within 3 days prior to study treatment and must agree to abstain from activities that could result in pregnancy from screening through 6 months after the last dose of study treatment, or patients of non-childbearing potential, where nonchildbearing potential is defined as follows (by other than medical reasons):

  * ≥45 years of age and has not had menses for >1 year;
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have levels of Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) in the post-menopausal range for women <50;
  * Post-hysterectomy, post-bilateral oophorectomy, or posttubal ligation: documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 6 months after the last dose of study treatment. Information must be captured appropriately within the site's source documents.
* 22. Female patients must agree not to breastfeed during the study and for 1 month after the last dose of study treatment.
* 23. Male patients whose partners are women of childbearing potential must use a condom during niraparib therapy and for 3 months after receiving the last dose of niraparib and must agree to abstain from activities that could result in pregnancy. In addition, men must not donate sperm during niraparib therapy and for 3 months after receiving the last dose of niraparib.

Exclusion Criteria:

* 1. HER2-positive disease based on local laboratory results (performed by IHC/in situ hybridization test) or unknown HER2 status.
* 2. Patients that are candidates for a local treatment with a radical intention.
* 3. Patients that have previously received any PARP inhibitor (PARPi), including niraparib, in metastatic setting. Note: Patients treated with PARPi on (neo)adjuvant regimen with disease-free interval greater than 24 months following treatment interruption are eligible.
* 4. Patients must not be simultaneously enrolled in any interventional clinical trial and must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
* 5. Patients who have had radiation therapy encompassing >20% of the bone marrow within 2 weeks prior to start of treatment, excepting for palliative radiation therapy to a small field >1 week prior to Day 1 of study.
* 6. Patients with visceral crisis who require chemotherapy.
* 7. Patients must not have a known hypersensitivity to niraparib components or excipients.
* 8. Patients must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
* 9. Patients must not have received colony-stimulating factors (e.g., Granulocyte colony-stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
* 10. Patients have had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy in adjuvant setting or cyclin-dependent kinases (CDK)4/6 inhibitors that persisted > 4 weeks and was related to the most recent treatment.
* 11. Patients must not have any known history of Myelodysplastic syndrome (MDS) or Acute myeloid leukemia (AML).
* 12. Patients must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (≤ 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan, any psychiatric disorder that prohibits obtaining informed consent, severe immunodeficiency disorders (i.e. human immunodeficiency virus [HIV] infection) or active hepatitis (i.e. Hepatitis B or C).
* 13. Patients must not have had diagnosis, detection, or treatment of another type of cancer ≤ 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin, cervical carcinoma in situ and ductal carcinoma in situ [DCIS] definitively treated).
* 14. PPatients with symptomatic uncontrolled brain metastases or leptomeningeal metastases. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression unless considered to have received definitive treatment for this condition and have evidence of clinically stable disease (SD) for 35 days.
* 15. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* 16. Patients who are unable to swallow orally administered medication.
* 17. Patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* 18. Chronic daily treatment with corticosteroids with a dose of ≥ 10 mg/day methylprednisolone equivalent (excluding inhaled steroids), except for prophylaxis use.
* 19. Female patients who are pregnant or breastfeeding, or adults of reproductive potential who are not using effective birth control methods.
* 20 .Patients unwilling to or unable to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) of niraparib in combination with AIs in unresectable locally advanced or metastatic HR-positive/HER2-negative breast cancer patients harboring either gBRCAms or gBRCAwt and HRD | Baseline up to 24 weeks
  The CBR as best response, defined as the percentage of patients who experience a complete response, partial response or stable disease for at least 24 weeks and assessed by modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) criteria

SECONDARY OUTCOMES:
Efficacy determinated by the Progression-free Survival (PFS) | Baseline up to 36 months
  PFS is defined as the time from the date of the first dose of study treatment until the first documented PD based on RECIST v1.1. or death due to any cause, whichever occurs first based on local investigator's assessment according to RECIST criteria v1.1.
Efficacy determinated by the Objective Response Rate (ORR) | Baseline up to 36 months
  The ORR is defined as the number of patients with CR and PR divided by the number of patients in the analysis set. Tumor response will be defined as best response based on local investigator's assessment according to RECIST criteria v.1.1.
Efficacy determined by Duration of Response (DoR) | Baseline up to 36 months
  DoR is defined as the time from first documented CR or PR until disease progression or death from any cause, based on local investigator's assessment according to RECIST criteria v1.1.
Efficacy determined by Overall survival (OS) | Baseline up to 36 months
  OS is defined as the time from the date of first dose of study treatment until death by any cause or the last date the patient was known to be alive.
Efficacy determined by Time to response (TTR) | Baseline up to 36 months
  Time to response (TTR) is defined as the time from the date of first dose of study treatment to the first objective tumor response observed for patients who achieved a Complete response (CR) or parcial response (PR).
Incidence of treatment-related AEs Grade 3 and 4 and serious adverse events (SAEs) [Safety] | Baseline up to 36 months
  Safety will be measured by using the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Llombart, Principal Investigator — MedSIR
Locations (10):
- Spain (10):
  - Centro Oncologico de Galicia, A Coruña
  - Complejo Asistencial de Ávila, Ávila
  - Hospital Uniersitario Vall d'Hebron, Barcelona
  - Hospital Clínic i provincial de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Instituto Valenciano de Oncología, Valencia

IPD SHARING:
Plan to Share IPD: No